CLINICAL TRIAL: NCT04672135
Title: A Phase 1 (First in Human) Randomized, Double-blind, Placebo-controlled SAD, MAD Study With an Adaptive Dose Design to Evaluate the Safety, Tolerability, and Pharmacokinetics of REM0046127 in Healthy Subjects
Brief Title: A Phase 1 (First in Human) Randomized, Double-blind, Placebo-controlled SAD, MAD Study With Oral REM0046127
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: reMYND (Industry)
Collaborators: NeuroScios GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: NSC20002
Record Dates: First submitted 2020-11-12; First posted 2020-12-17 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: A Single Ascending Dose study with 6 Cohorts with 8 young male subjects each and 1 cohort with 4 male and 4 female subjects A Multiple Ascending Dose MAD study with 2 Cohorts: (Cohort 1: 10 young male subjects, Cohort 2: 6 elderly male and 6 elderly female (not of CBP) subjects.
Who Masked: Participant, Investigator
Masking Description: An independent statistician will provide the randomization list to an unblinded person at the site. The unblinded person prepares the medication for the subjects. The ready medication is handed over to the blinded investigator and the investigator will dose the blinded subjects.
  Randomization numbers will be kept secret until data base lock. After data base lock the results will be unblinded for final analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Drug (Active Comparator): Each subject receives either a single dose (SAD) or a multiple dose (MAD) of REM0046127 as oral solution with a concentration of 100 mg/mL REM0046127. The starting dose for the first cohort in the SAD is 35mg up to a maximum of 2000mg at cohort 5. The starting dose for the MAD study is 0,75 of the Maximum Tolerated Dose (MTD) from the SAD.
  Interventions: Drug: REM0046127
- Placebo (Placebo Comparator): Each subject receives either a single (SAD) or multiple (MAD) dose of REM0046127 as oral solution with a concentration of 0 mg/mL REM0046127. The dose for each cohort is corresponding the amount of solution needed in the verum group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REM0046127 — Oral solution: 100 mg/mL REM0046127
  Arms: Study Drug
Drug: Placebo — Oral solution with 0 mg/mL REM0046127
  Arms: Placebo

SUMMARY:
This is a phase 1 randomized double blind, first in human (FIH) study with the novel oral Alzheimer drug candidate REM0046127, which consists of two main parts, a single ascending dose (SAD) study with 7 cohorts followed by a multiple ascending dose (MAD) study with 2 cohorts.

DETAILED DESCRIPTION:
SAD

As a baseline, 5 cohorts of 8 young healthy males are foreseen, with a repeat to assess food impact and an additional elderly cohort. Depending on the early FIH findings, the number of cohorts could be more or less. FIH studies include initially only males due to the incomplete nature of preclinical reproductive toxicology studies

* Treatment duration: single day
* Each cohort:

  * 2 volunteers on placebos, of which 1 sentinel
  * 6 volunteers on study drug, of which 1 sentinel
* Timing for each cohort will be about 21 days

  * Subjects will be screened for selection from day -21 to day -1 before starting the experimental phase of each cohort
  * First the 2 sentinels will be dosed
  * Following the review of sentinel safety and tolerability data through the Data Safety Monitoring Board (DSMB) after one day or 2 half-life times following the sentinel dosing, the remaining 1+5 subjects will be randomized and dosed approximately 7 days after the sentinels

MAD

* First cohort of 10 healthy young male subjects. This cohort can be initiated after the food interaction has been assessed in the last safe SAD cohort, and does not need to wait for the elderly cohort.
* Second cohort of 12 healthy elderly subjects:

  * The 1st cohort of healthy young male at about 75% of the Maximum Tolerated Dose (MTD) of the SAD
  * The 2nd cohort of healthy older male and female (not of child-bearing potential) at about 50 or 100% of the highest tolerable dose of the SAD, depending on the observations in the 1st MAD cohort to assess potential impact of age on Pharmacokinetics (PK)
  * Treatment duration: 7 days
  * Timing for each cohort will be about 35 days
* Subjects will be screened for selection from day -21 to day -1 before starting the experimental phase each cohort
* First the sentinels will be dosed
* Following the review of sentinel safety and tolerability data through the DSMB, the remaining subjects will be randomized and dosed approximately 14 days later
* According to plan the sentinels of the 2nd cohort will be dosed about 35 days after the sentinels of the 1st cohort.

ELIGIBILITY:
Inclusion Criteria:

1. SAD/MAD: Young male subjects aged 18 to 45 years (limits included) willing and able to give their written consent to participate in the trial after having received information about the study design, the objectives of the project, the possible derivative risks, and their right to withdraw from the study at any time and for any reason
2. Elderly Cohorts: Elderly male and female (not of childbearing potential) subjects aged 55 to 80 (limits included) willing and able to give their written consent to participate in the trial after having received information about the study design, the objectives of the project, the possible derivative risks, and their right to withdraw from the study at any time and for any reason.
3. Women not of childbearing potential: Clinically significant abnormalities in screening laboratory tests, including:

   * Surgically sterile (bilateral tubal ligation, hysterectomy), or
   * Postmenopausal with last natural menses greater than 24 months
4. Electrocardiogram without clinically significant pathologic abnormalities and with corrected QT interval (cQT) values lesser than 450 ms
5. Normotensive as defined by Systolic Blood Pressure ≤ 150 mm Hg. Diastolic Blood Pressure ≤ 90 mm Hg without antihypertensive medication
6. Body Mass Index (BMI) between 18 and 30 kg/m2.
7. Body weight between 60 and 80 kg, inclusive

   Only for the elderly cohort of the MAD:
8. Participants may be taking medication for non-serious chronic diseases, provided that the dose of these concomitant medications has been stable within the previous 2 months
9. No suicidal ideation, as demonstrated by a score of "0" on the Columbia Suicide Severity Rating Scale (C-SSRS)

Exclusion Criteria:

1. Women of childbearing potential (WOCBP)
2. Failure to perform screening or baseline examinations
3. Any chronic medical condition (such as type 1 diabetes) requiring chronic treatment that might increase the risk to the subject or confound the interpretation of safety observations according to the clinical assessment of the investigator (physician)
4. Evidence of active infection requiring antibiotic therapy within 14 days prior to screening
5. Medical history of vasculitis or any autoimmune disease excluding seasonal allergic rhinitis and childhood history of atopic dermatitis
6. History of any treatment for cancer within the past 2 years, other than basal cell or squamous cell carcinoma of the skin
7. Seropositive for human immunodeficiency virus (HIV)
8. History of acute/chronic hepatitis B or C and/or carriers of hepatitis B (seropositive for Hepatitis B surface antigen [HbsAg] or anti-Hepatitis C [Hepatitis C Virus (HCV)] antibody)
9. Clinically significant abnormalities in screening laboratory tests, including:

   * Absolute neutrophil count < 1.4 x109
   * Absolute lymphocyte count < 1.2 x 109
   * Alanine transaminase (ALT) or aspartate transaminase (AST) > 1.5 x the upper limit of normal (ULN)
   * Lactate Dehydrogenase (LDH) > 1.5 x ULN
   * Total bilirubin level: Out of normal range 0-1.5 mg/dL
   * Estimated glomerular filtration rate (eGFR) < 60 mL/min
   * Haemoglobin (Hgb): out of normal range (male: 13,5-18,0 g/dL).
   * Haemoglobin (Hgb): out of normal range (female: 12,0-16,0 g/dL)
10. Use of an investigational drug within 2 months prior to dosing in this study
11. Any disorder that could interfere with the absorption, distribution, metabolism or excretion of drugs (e.g. small bowel disease, Crohn's disease, celiac disease, or liver disease)
12. Chronic kidney disease (defined as the presence of any degree of proteinuria on urine analysis and/or an eGFR of <60 ml/min using the (Modification of Diet in Renal Disease (MDRD) formula)
13. Psychiatric history of current or past psychosis, bi-polar disorder, major depression, or anxiety disorder requiring chronic medication within the past 5 years
14. History of substance abuse, including alcohol and nicotine or positive urine drug screen at screening visit
15. Any reason or opinion of the investigator that would prevent the subject from participation in the study
16. Inability to follow the instructions or an unwillingness to collaborate during the study
17. Male subjects with female partner of child-bearing potential who are unwilling or unable to adhere to contraception requirements

    Only for the elderly cohort of the MAD:
18. Chronic daily drug intake during the study period:

    * Benzodiazepines, neuroleptics or major sedatives
    * Antiepileptics
    * Centrally active anti-hypertensive drugs (clonidine, l-methyl-DOPA, guanidine, guanfacine, etc.)
    * Opioid containing analgesics
19. History of cancer within the last 5 years, except basal cell carcinoma, non-squamous skin carcinoma, prostate cancer or carcinoma in situ with no significant progression over the past 2 years
20. Clinically significant, advanced or unstable disease that may interfere with primary or secondary variable evaluations, and which may bias the assessment of the clinical or mental status of the volunteer or put the volunteer at special risk, such as:

    * Chronic liver disease, liver function test abnormalities or other signs of hepatic insufficiency (Alanine-Aminotransferase (ALT), Aspartate-Aminotransferase (AST), Gamma Glutamyl-Transferase (GT), alkaline phosphatase > 2.0 ULN)
    * Respiratory insufficiency
    * Heart disease (myocardial infarction, unstable angina, heart failure, cardiomyopathy within six months before screening)
    * Bradycardia (heartbeat <50/min) or tachycardia (heartbeat >95/min)
    * Hypertension (<180/95) or hypotension requiring treatment with more than 2 drugs
    * Atrioventricular (AV) block (type II / Mobitz II and type III), congenital long QT syndrome, sinus node dysfunction or prolonged QTcF-interval (males >450 and females >470 ms)
    * Uncontrolled diabetes defined by HbA1c >8.5
    * Renal insufficiency (serum creatinine > 2mg/dL) or creatinine clearance ≤ 30 mL/min according to Cockcroft-Gault formula).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-26 (Actual)

PRIMARY OUTCOMES:
Adverse Events | SAD: from dosing to 72 hours after dosing. MAD: from the first dosing until 48 hours after the last dosing on day 7.
  Number of Adverse Events either related or not related to treatment in the verum group in comparison to the placebo group
SAD: Plasma Concentration including Peak Plasma Concentration (Cmax) | Plasma samples will be taken during SAD at baseline and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose.
  The plasma concentration during 48 hours after the dosing.
SAD: Plasma Concentration including Half-Life(t1/2) | Plasma samples will be taken during SAD at baseline and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose.
  The plasma concentration during 48 hours after the dosing.
SAD: Area under the Curve (AUC) | Plasma samples will be taken during SAD at baseline and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 18, 24, 36 and 48 hours post-dose.
  The AUC between baseline and 48 hour safter dosing.
MAD: Half-Life(t1/2) between Baseline and 48 hours after the last dosing. | Plasma samples will be taken pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 hours post-dose, pre-dose on Day 5 and on Day 7: 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 hours (Day 8) and 48 hours (Day 9).
  Half-Life(t1/2) between Baseline and 48 hours after the last dosing.
MAD: Plasma Concentration | Plasma samples will be taken pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 hours post-dose, pre-dose on Day 5 and on Day 7: 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 hours (Day 8) and 48 hours (Day 9).
  Peak Plasma Concentration (Cmax) between Baseline and 48 hours after the last dosing.
MAD: Area under the Curve (AUC) | Plasma samples will be taken pre-dose and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 hours post-dose, pre-dose on Day 5 and on Day 7: 0, 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24 hours (Day 8) and 48 hours (Day 9).
  The AUC and steady-state volume of distribution(Vss) during the time interval from the first dose and 48 hour safterlast dose
Cerebrospinal Fluid (CSF) PK (MAD) | CSF samples will be collected on the last day of dosing (Day 7) at approximately Tmax determined during SAD
  In CSF the unbound brain/plasma partition coefficient (Kp,u) will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Nikola Helmberg, PhD, Study Director — NeuroScios GmbH
Locations (1):
- Medical University Vienna, Department of Clinical Pharmacology, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No